CLINICAL TRIAL: NCT04114331
Title: Feasibility of a Post-Hospitalization PT Intervention in Patients With Pneumonia
Brief Title: Feasibility of a Physical Therapy Intervention on Older Adults With Hyperkyphosis or Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0098
Record Dates: First submitted 2019-09-16; First posted 2019-10-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-08

CONDITIONS: Pneumonia; COPD; Hyperkyphosis; Postural, Thoracic Kyphosis
Keywords: forward head posture
MeSH Terms: conditions — Pneumonia; Pulmonary Disease, Chronic Obstructive; Kyphosis | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual therapy and exercise (Experimental): The intervention (3 times a week for 4 weeks, for a total of 12 sessions) consisted primarily of manual therapy (soft tissue and joint mobilization) followed by therapeutic exercises (muscular control and coordination).
  Manual therapy:
  Joint mobilizations (Grades I-V) to cervical spine, thoracic spine and ribs Soft tissue mobilization to the pectoralis, scaleni, upper traps, thoracolumbar fascia, erector spinae, and suboccipital musculature
  Therapeutic exercises:
  Strengthening of mid and lower traps, lats, glut med, and glut max. Active & passive stretching of thoracic and lumbar rotation, hip flexors, and plantarflexors.
  The treating therapists agreed on a protocol with treatment individualized to each patient.
  Interventions: Other: Manual therapy and exercise

INTERVENTIONS:
Other: Manual therapy and exercise — Manual therapy consisting of soft tissue and joint mobilization to gain mobility. Therapeutic exercise was active motion and resisted motion to gain motor control and motor coordination in the new range.

SUMMARY:
The original intent was to use a manual therapy and therapeutic exercise intervention with older patients with pneumonia post-hospitalization. It was hypothesized that the physical therapy intervention would have a positive impact on posture, physical function, pulmonary function, gait, quality of life, and ultimately readmission. This patient population was found to be not feasible to recruit and the study target population was expanded to include older community dwelling adults with pneumonia, chronic obstructive pulmonary disease (COPD), or hyperkyphosis.

DETAILED DESCRIPTION:
This original study was a feasibility study to determine the ability to recruit and to assess pilot data to determine the effects of a physical therapy intervention on physical function, gait, balance, posture, pulmonary function, and quality of life. Additionally the 30 day readmission, ER visits, and mortality was to be tracked. This study failed due to lack of recruitment. However, the aim to examine the effectiveness a physical therapy intervention was still used just in a broader population. The intervention and measures remained the same except for 30 day admission/mortality data.

The new aim was to examine the effectiveness of manual therapy and exercise on posture, function, gait, pulmonary function, and quality of life in older community dwelling adults with hyperkyphosis or forward head posture. Kyphosis, osteoporosis, decreased trunk flexibility, and pain are considered potential causes of restrictive lung function. The physical therapy intervention targets both soft tissue and skeletal restrictions to improve mobility. The outcomes were chosen to examine not only the direct impact on posture but also the indirect impact on physical function including pulmonary status. Lastly, cognitive mapping was used to record the change in the perceptions of the participants as they improved.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years of age
* hyperkyphosis, forward head posture, pneumonia, or chronic obstructive pulmonary disease (COPD)
* community dwelling
* self report of ability to walk 10 feet or greater with or without an assistive device
* ability to perform informed consent
* ability to transport to research facility
* ability to read and write in English or Spanish

Exclusion Criteria:

* Inability to perform informed consent
* Inability to follow directions
* Inability to perform transfers, sit, and stand independently
* Inability to ambulate 10 feet or more with or without an assistive device
* Inability to perform pulmonary function testing
* Inability to fully participate in testing and measures
* Inability to fully participate in the intervention
* Severe claustrophobia
* Unable to tolerate physical touch
* Morbid obesity (BMI greater than 40)
* History of prior lung disease such as cancer or transplant
* History of comorbidity that would affect lung function such as neuromuscular disease (ALS, MS), collagen disease (SLE), cardiovascular disease (CHF), or musculoskeletal disease with an autoimmune component (Ankylosing Spondylosis, RA).
* A prior discharge within 30 days of hospitalization for pneumonia or COPD
* Discharge against medical advice

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Posture, as measured by change in height | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Height in cm
Posture, as measured by change in kyphotic index | through study completion (4 weeks) and one time follow-up at an average of 6 months
  kyphotic index = (thoracic width/thoracic height) *100 as measured from flexicurve tracing. A flexible ruler is molded to the posterior spine from C7 to the lumbosacral interspace. Ruler is placed on paper and traced. Measures of the thoracic width and height are taken in centimeters.
Posture, as measured by change in block test | through study completion (4 weeks) and one time follow-up at an average of 6 months
  height of blocks (measured in cm) under the head with participant supine
Posture, visual change in digital photos | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Digital photo in standing anterior and side views as well as supine view

SECONDARY OUTCOMES:
Function as a change in Timed Up and Go speed | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Timed Up and Go as measured in seconds to performed standardized functional test. Participants are timed in seconds from sitting in a chair to standing, walking 3 meters, turning around, walking back, and sitting down.
Function as a change in Functional Reach test | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Functional reach as measured in cm. It is performed by having the participant standing still and is instructed to reach forward as far as you can without taking a step.
Function as a change in the Short Physical Performance Battery (SPPB) score | through study completion (4 weeks) and one time follow-up at an average of 6 months
  SPPB score as determined by seconds to perform each component of this standardized test. This functional test has 3 components of 5 times sit to stand, gait speed, and balance. 5 times sit to stand is a standardized test of lower extremity strength that is performed by rising and sitting in a chair 5 times in a row. The activity is timed. Gait speed will be extracted from gaitrite data. Balance tests will be timed.
Function and Gait as a change in the 2 Minute Walk Test (2MWT) | through study completion (4 weeks) and one time follow-up at an average of 6 months
  2MWT is the measured as the distance (feet) covered in 2 minutes
Function and patient perception as change in the Patient Specific Functional Scale (PSFS) | through study completion (4 weeks) and one time follow-up at an average of 6 months
  PSFS is a standardized survey of activities that are difficult to perform (listed by participant) and to what degree as measured on a likert scale (0 to 10)
Gait as measured by change in gait parameters on a Gaitrite walkway | through study completion (4 weeks) and one time follow-up at an average of 6 months
  The gaitrite records a standard set of parameters. Change in gait speed (m/sec), step length (cm), stride length (cm), double limb support time (seconds), and step width (cm)
Gait as measured by change in Tekscan measures of force | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Tekscan records a standard set of measures of time and force. Change in peak force at loading response, mid-stance, and terminal stance in newtons.
Pulmonary function change measure by spirometry | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Spirometry provides standard measures of respiratory volume and volume in time. Changes in Forced Vital Capacity and Forced Expiratory Volume in 1 second were the measures of interest.
Patient perception as measured by changes in Cognitive Mapping | through study completion (4 weeks) and one time follow-up at an average of 6 months
  Cognitive mapping provides the issues, concerns, and perceptions of the participants of how posture affects their life. Measured by words recorded and qualitative analysis.

OTHER OUTCOMES:
Weight | through study completion (4 weeks) and one time follow-up at an average of 6 months
  measured in pounds

CONTACTS AND LOCATIONS:
Overall Officials: Lynne C Hughes, PhD, PT, Principal Investigator — University of Texas
Locations (1):
- School of Health Professions at the University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Hughes LC, Ellis AL, Rogers HL, Hadley M, Galloway RV. A secondary analysis of gait after a 4-week postural intervention for older adults with hyperkyphosis. BMC Musculoskelet Disord. 2025 Feb 11;26(1):136. doi: 10.1186/s12891-025-08330-7. PMID 39934800
- [Derived] Hughes LC, Galloway RV, Fisher SR. Feasibility of a 4-Week Manual Therapy and Exercise Intervention on Posture and Function in Community-Dwelling Older Adults: A Pilot Study. J Geriatr Phys Ther. 2022 Jul-Sep 01;46(3):151-160. doi: 10.1519/JPT.0000000000000360. Epub 2022 Aug 5. PMID 35939663